CLINICAL TRIAL: NCT03414645
Title: Randomized Multicenter Double-Masked Placebo-Controlled Parallel Phase I/II Study to Determine the Safety and Exploratory Efficacy of Topical Fibrinogen Depleted Human Platelet Lysate in Patients With Dry Eye Secondary to Graft vs Host Disease
Brief Title: Topical Fibrinogen-Depleted Human Platelet Lysate in Patients With Dry Eye Secondary to Graft vs. Host Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cambium Bio Limited (Industry)
Collaborators: Massachusetts Eye and Ear Infirmary (Other); Oregon Health and Science University (Other); University of Michigan (Other); Duke University (Other); Stanford University (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAM-101
Record Dates: First submitted 2018-01-08; First posted 2018-01-30 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Dry Eye; Graft-versus-host-disease; Ocular Discomfort
MeSH Terms: conditions — Dry Eye Syndromes; Graft vs Host Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CAM-101 10% (Experimental): FD hPL 10 vol/vol %
  Interventions: Biological: CAM-101 10%
- CAM-101 30% (Experimental): FD hPL 30 vol/vol %
  Interventions: Biological: CAM-101 30%
- Vehicle Control (Placebo Comparator): PlasmaLyte-A, vehicle control, a preservative-free ophthalmic drop
  Interventions: Biological: Vehicle Control

INTERVENTIONS:
Biological: CAM-101 10% — fibrinogen-depleted human platelet lysate
  Other Names: FD hPL 10% vol/vol
  Arms: CAM-101 10%
Biological: Vehicle Control — PlasmaLyte-A, vehicle control, a preservative-free ophthalmic drop
  Arms: Vehicle Control
Biological: CAM-101 30% — fibrinogen-depleted human platelet lysate
  Other Names: FD hPL 30% vol/vol
  Arms: CAM-101 30%

SUMMARY:
The purpose of this Phase 1/2 study is to compare the safety and tolerability of four times a day (QID) dosing of a non-preserved topical ocular drop formulation of 10 vol/vol % and 30 vol/vol % of FD hPL to vehicle control eye drops in patients with Dry Eye Disease (DED) secondary to Graft vs. Host Disease (GvHD).

DETAILED DESCRIPTION:
For patients who do not find relief from other modes of therapy, autologous serum tears have been used as an alternative therapy since the mid-1980s. Limitations such as the need for periodic blood draws, the lack of standardization in the preparation of AST and platelet-enriched plasma tears, the unknown shelf life of AST preparations, the use of non-preserved multi-dose packaging and the practical difficulties patients face in storing these products frozen or refrigerated have hindered their widespread use for treating GvHD and other forms of severe tear deficiency.

To address these shortcomings, Cambium Medical Technologies, LLC has developed a proprietary method of standardizing and manufacturing a fibrinogen-depleted standardized platelet lysate using pooled human platelet lysates (phPL) collected from qualified healthy donors (CAM-101). Because Cambium's proprietary manufacturing process depletes pooled human platelet lysates of fibrinogen (the key clotting protein in platelets), the remaining product contains enriched levels of several key nutritive and regenerative components than are normally found in non-standardized AST as well as healthy tear film.

Given the multi-factorial nature of DED, the enriched levels of numerous key nutritive components in CAM-101 may well prove to be superior to artificial tears and certain single active ingredient products which treat only one cause or contributor of dry eye (e.g., inflammation) and other forms of tear deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, of age 18 years (inclusive) or older at the time of signing the ICF;
2. Diagnosis of DED secondary to GvHD following allogeneic hematopoietic stem cell transplantation as determined by medical history
3. For females:

   1. Be of non-child-bearing potential. Surgically sterilized (e.g., hysterectomy or bilateral oophorectomy) for at least 6 months prior to screening or postmenopausal (postmenopausal women must have no menstrual bleeding for at least 1 year prior to screening) and menopause will be confirmed by a plasma FSH level of >40 IU/L) or
   2. Women of childbearing potential must be non-lactating and agree to use a highly effective acceptable form of birth control (e.g., established hormonal birth control plus a barrier method, double barrier method: intrauterine device plus condom or spermicidal gel plus condom) from 21 days prior to dosing until 7 days after dosing, and
   3. Women with a negative pregnancy test (β-hCG assay) in urine at screening and Day 1 predose;
4. Schirmer tear test with anesthesia <7 mm/5 min in at least one eye during screening;
5. Willingness and and ability to undergo, and return for, all scheduled study-related visits through Follow-up;
6. Willingness and and ability to provide written Informed Consent consistent with privacy language as per national regulations (e.g., HIPAA authorization) and which signature may be obtained from the patient or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication);
7. Willingness to communicate with the Investigator and site staff and comply with all study procedures and requirements;
8. Agreement not to participate in another interventional study while participating in this study.

Exclusion Criteria:

1. Any abnormal lid anatomy or blinking function in either eye;
2. Any history of other ocular disease requiring topical ocular treatment other than artificial tears and/or Restasis® (cyclosporine ophthalmic emulsion; Allergan Irvine, CA) or Xiidra® (lifitegrast, Shire, Lexington, MA). Patients currently using Restasis® or Xiidra® for conditions other than DED (e.g., allergies);
3. Previous intraocular or ocular laser surgery within the past 3 months or any refractive surgery procedure within the past 6 months of the screening visit in either eye;
4. Any relevant ocular anomaly interfering with the ocular surface, including active ocular herpes simplex infection, recurrent corneal erosion, symptomatic epithelial basement membrane dystrophy, mucus fishing syndrome, giant papillary conjunctivitis, post-radiation keratitis, Stevens-Johnson syndrome, corneal ulcer, abnormalities of the nasolachrymal drainage system, chemical injury, destruction of the conjunctival goblet cells or scaring, diagnosed significant anterior blepharitis and/or progressive pterygium, or any other additional condition(s) associated with or causing dry eye;
5. Presence or history of any ocular disorder or condition, including ocular surgery (including palpebral and cataract surgery, trauma), infection (viral, bacterial, fungal), disease or inflammation not associated with dry eye unless disorder or disease is:

   1. Stable for at least 3 months before the Screening Visit; and
   2. As determined by the Investigator not likely to impact or possibly interfere with the interpretation of study results.
6. History of ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis other than dry eye;
7. Known hypersensitivity to one of the components of the study or procedural medications (e.g., fluorescein, lissamine green, Refresh Plus®);
8. Inability to refrain from contact lens wear during the study, including the 2 week Run-in period;
9. Anticipated temporary or permanent need for punctal plugs during the study, except if punctal plugs have been in place for at least 2 weeks prior to Screening, in which case the plugs are allowed to remain in place during the study; if plugs should fall out during the course of the study, the instance will be recorded and the plug(s) can be replaced;
10. Ocular or clinically significant systemic disease (e.g., diabetes with glycemia out of range, thyroid malfunction, uncontrolled autoimmune disease) or condition(s) not stabilized within 1 month (30 days) before Screening or a condition judged by the Investigator to be incompatible or interferes with the study results;
11. Inability or unwillingness to discontinue use of autologous or platelet rich plasma eye drops during the 2 week washout period and the duration of the study;
12. Anticipated change in the use or dose of Restasis®, Xiidra®, or artificial tears within 14 days before Screening or during the study. If currently taking Restasis®, Xiidra®, or artificial tears, treatment(s) for DED can continue throughout the study without a change in dose. If currently using Restasis® or Xiidra® for conditions other than DED, then patient will be excluded from study. If not currently taking Restasis®, Xiidra® or artificial tears, these drugs cannot begin during the study;
13. Anticipated change in the patient's use of or dosage of systemic medications that could affect tear function (e.g., antihistamines, tricyclic antidepressants, anxiolytics, antimuscarinics, beta-blocking agents, phenothiazines, tacrolimus, sirolimus, etc.) during the study. If currently taking any of these drugs, treatment(s) can continue throughout the study without a change in dose;
14. Pregnancy or breast feeding at the time of study entry;
15. History of clinically significant drug or food allergy;
16. Positive HIV, hepatitis B or C viral test at screening;
17. History, as judged by the Investigator, of drug or alcohol abuse (i.e., alcohol consumption >2 drinks/day over the last 3 months prior to screening); drug abuse is any use of illegal drugs or prescription-drug over usage or addiction;
18. Taken any investigational medication and/or participated in any clinical studies within 30 days of screening;
19. Any patient who, in the judgment of the Investigator, may not be able to cooperate fully with the study staff, may have difficulty following some study requirements, or is otherwise not qualified for the study;
20. Any patient who is directly involved in the conduct of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with ocular treatment-related adverse events as assessed by CTCAE v4.0 | 42 Days
  To evaluate the safety and tolerability of two concentrations of CAM-101 (FD hPL 10 vol/vol % and 30 vol/vol %) topical ophthalmic solution in patients with dry eye disease (DED) secondary to graft versus host disease (GvHD) after 6 weeks (42 days) of treatment.
  The primary outcome measure:
  Percentage of patients in each dose group with ocular adverse events at Day 42
Number of participants with systemic treatment-related adverse events as assessed by CTCAE v4.0 | 42 Days
  Number of participants with ocular treatment-related adverse events as assessed by CTCAE v4.0 To evaluate the safety and tolerability of two concentrations of CAM-101 (FD hPL 10 vol/vol % and 30 vol/vol %) topical ophthalmic solution in patients with dry eye disease (DED) secondary to graft versus host disease (GvHD) after 6 weeks (42 days) of treatment.
  The primary outcome measure:
  Percentage of patients in each dose group with systemic adverse event at Day 42
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 42 Days
  To evaluate the safety and tolerability of two concentrations of CAM-101 (FD hPL 10 vol/vol % and 30 vol/vol %) topical ophthalmic solution in patients with dry eye disease (DED) secondary to graft versus host disease (GvHD) after 6 weeks (42 days) of treatment.
  The primary outcome measure:
  The percentage of patients in each dose group that show a change from Normal to Abnormal with clinical significance in any ocular examination assessment at Day 42

SECONDARY OUTCOMES:
Efficacy as measured by change in corneal staining | 42 Days
  To evaluate the preliminary efficacy of two concentrations of FD hPL (10 vol/vol % and 30 vol/vol %) to each other and to a vehicle control in the treatment of patients with DED secondary to GvHD as the result of allogeneic stem cell transplantation as measured by change in corneal staining:
  * Change from baseline in fluorescein corneal staining on Day 42
  * Change from baseline in lissamine green corneal staining on Day 42
Efficacy as measured by ocular surface disease index (OSDI) | 42 Days
  To evaluate the preliminary efficacy of two concentrations of FD hPL (10 vol/vol % and 30 vol/vol %) to each other and to a vehicle control in the treatment of patients with DED secondary to GvHD as the result of allogeneic stem cell transplantation as measured by ocular surface disease index (OSDI)
  Change from baseline in OSDI score on Day 42
  o The OSDI is assessed on a scale of 1-100 with higher scores representing greater disability The OSDI questionnaire includes total, visual-related function, and trigger subscales The Index is determined by multiplying the sum of the scores from each question by 25 and dividing the product by the number of questions answered.
  A continuum of scores from normal to dry has been developed
Efficacy as measured by ocular discomfort using the 100 point visual analogue scale (VAS) scores | 42 Days
  To evaluate the preliminary efficacy of two concentrations of FD hPL (10 vol/vol % and 30 vol/vol %) to each other and to a vehicle control in the treatment of patients with DED secondary to GvHD as the result of allogeneic stem cell transplantation as measured by ocular discomfort using the 100 point visual analogue scale (VAS) scores
  Change from baseline in ocular discomfort score as measured with VAS on Day 42VAS Patients will be asked questions about their current ocular discomfort by indicating from 0 (no discomfort) to 100 (maximal discomfort)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Waller, MD PhD, Study Director — Cambium Bio Limited
Locations (6):
- United States (6):
  - Byers Eye Institute of Stanford University, Palo Alto, California
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Michigan - Kellogg Clinical Research Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University Eye Center, Durham, North Carolina
  - Oregon Health Sciences University - Casey Eye Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No